CLINICAL TRIAL: NCT01513733
Title: The CATCH Prostate Cancer Trial: Cabazitaxel And Tasquinimod in Men With Castration-Resistant Heavily Pre-treated Prostate Cancer
Brief Title: The CATCH Prostate Cancer Trial: Cabazitaxel And Tasquinimod in Men With Prostate Cancer
Acronym: CATCH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew J. Armstrong, MD (Other)
Responsible Party: Sponsor-Investigator, Andrew J. Armstrong, MD, Assoc Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00032421; c11-082 (Other Grant/Funding Number: PCCTC)
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — tasquinimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tasquinimod single dose (Experimental)
  Interventions: Drug: tasquinimod
- tasquinimod 0.25 mg followed by 0.5 mg (Experimental): tasquinimod 0.25 mg for 3 weeks followed by 0.5 mg continuously, if tolerated
  Interventions: Drug: tasquinimod 0.25 mg; 0.5 mg
- tasquinimod 0.25 mg; 0.5 mg; 1.0 mg (Experimental): tasquinimod 0.25 mg for 3 weeks followed by 0.5 mg for 3 weeks followed by 1.0 mg continuously, if tolerated
  Interventions: Drug: tasquinimod 0.25 mg; 0.5 mg; 1.0 mg

INTERVENTIONS:
Drug: tasquinimod — tasquinimod 0.25 mg continuously
  Arms: Tasquinimod single dose
Drug: tasquinimod 0.25 mg; 0.5 mg — tasquinimod 0.25 mg for 3 weeks followed by 0.5 mg continuously, if tolerated
  Arms: tasquinimod 0.25 mg followed by 0.5 mg
Drug: tasquinimod 0.25 mg; 0.5 mg; 1.0 mg — tasquinimod 0.25 mg for 3 weeks followed by 0.5 mg for 3 weeks followed by 1.0 mg continuously, if tolerated
  Arms: tasquinimod 0.25 mg; 0.5 mg; 1.0 mg

SUMMARY:
The standard of care for men with metastatic CRPC in 2010 following progression on docetaxel is cabazitaxel or abiraterone acetate/prednisone. Based on results from two other studies, cabazitaxel and prednisone has become a standard second line chemotherapy regimen and becomes the backbone upon which to improve upon. Thus, the primary objective of this study is to determine the recommended dose of tasquinimod in combination with cabazitaxel and prednisone based on safety and tolerability in men with chemorefractory metastatic castration-resistant prostate cancer (CRPC).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the prostate without small cell features;
2. At least 18 years of age when signing the Informed Consent;
3. Presence of metastatic disease on bone scan or CT/MRI imaging;
4. Ongoing androgen deprivation therapy with a gonadotropin releasing hormone (GnRH) analogue or orchiectomy (i.e., medical or surgical castration);
5. For patients who have not had an orchiectomy, there must be a plan to maintain effective GnRH-analogue therapy for the duration of the trial;
6. Serum testosterone level < 50 ng/dL at the Screening Visit;
7. Progressive disease on or following docetaxel-based chemotherapy with medical or surgical castration. Patients who are intolerant of docetaxel are also allowed. Disease progression for study entry is defined as one or more of the following three criteria: 1) PSA progression defined by a minimum of three rising PSA levels with an interval of ≥ 1 week between each determination. The PSA value at the Screening visit should be ≥ 2 μg/L (2 ng/mL); 2) Soft tissue disease progression defined by RECIST 1.1; 3) Bone metastatic disease progression defined by one or more new lesions on bone scan that are not clinically consistent with tumor flare;
8. No more than three prior chemotherapy regimens with at least one regimen containing docetaxel (unless intolerant as per # 7 above);
9. Karnofsky Performance Status of >70;
10. Estimated life expectancy of at least three months;
11. Able to swallow the study drug and comply with study requirements;
12. Willing and able to give informed consent.

Exclusion Criteria:

1. Subjects > 80 years old (dose escalation phase only, due to lower clearance in elderly patients);
2. Severe concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment;
3. Metastases in the brain or active epidural disease (NOTE: patients with treated epidural disease are allowed provided follow up imaging documents stability of epidural disease);
4. Absolute neutrophil count < 1,200/μL, platelet count < 100,000/μL, and hemoglobin <9 g/dL at the Screening Visit; (NOTE: patients may not have received any growth factors or blood transfusions within seven days of the hematologic laboratory values obtained at the Screening Visit)
5. Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 times the upper limit of normal at the Screening Visit;
6. Creatinine > 1.5 x ULN at the Screening visit;
7. History of another malignancy within the previous 3 years other than non-melanomatous skin cancer or non-invasive bladder cancer treated with curative intent;
8. Treatment with androgen receptor antagonists (bicalutamide, flutamide, nilutamide, MDV3100), 5-α reductase inhibitors (finasteride, dutasteride), estrogens (ie DES), sipuleucel-T, or chemotherapy within 28 days of Day 1 visit or plans to initiate treatment with any of these treatments during the study;
9. Use of herbal products that may decrease PSA levels or systemic corticosteroids greater than the equivalent of 10 mg of prednisone/prednisolone per day within four weeks of Day 1 visit;
10. Ongoing treatment with warfarin unless the international normalized ratio (INR) is well controlled and below 4
11. Exposure to ketoconazole or other strong CYP3A4 inhibitors or inducers intravenously or orally within 28 days prior to Day 1 Visit. For abiraterone acetate or TAK700, 14 days washout is needed.
12. Ongoing treatment with sensitive CYP1A2 substrates or CYP1A2 substrates with narrow therapeutic range (Appendix 3).
13. Ongoing treatment with CYP3A4 substrates with narrow therapeutic range (Appendix 3).
14. Radiation therapy within 2 weeks (if single fraction of radiotherapy within 2 weeks) and radionuclide therapy within 8 weeks of Day 1 visit;
15. Planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery;
16. Structurally unstable bone lesions suggesting impending fracture;
17. Clinically significant cardiovascular disease including:myocardial infarction within 6 months, uncontrolled angina within 3 months, congestive heart failure, Diagnosed or suspected congenital long QT syndrome; significant ventricular arrhythmias, Prolonged corrected QT interval by the Fridericia or Bazett correction formula, History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place; Hypotension (systolic blood pressure < 86 mMHg or bradycardia with a heart rate < 50 beats per minute on any ECG taken at the Screening or Day 1 visit; Uncontrolled hypertension; TIA or stroke/CVA within 6 months of Day 1 visit; Rest limb claudication or ischemia within 6 months of Day 1 visit
18. Use of an investigational agent within four weeks of Day 1 visit or plans to initiate treatment with an investigational agent during the study;
19. Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last three months);
20. Major surgery within four weeks prior to Day 1 visit.
21. Presence of NCI CTC grade >1 peripheral neuropathy
22. History of pancreatitis
23. Known positive serology for HIV (patients with known history of HIV will be excluded because of potential for unforeseen toxicity and morbidity in an immunocompromised host).
24. Chronic hepatitis B or C with advanced, decompensated hepatic disease, or cirrhosis of the liver or history of a chronic viral hepatitis or known viral hepatitis carrier (patients recovered from hepatitis will be allowed to enter the study).
25. Documented prior disease progression on tasquinimod -

Ages: 18 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience dose limiting toxicities at the highest titrated dose for each dose level | 6 weeks
  The primary objective is to determine the recommended dose of tasquinimod in combination with cabazitaxel and prednisone based on safety and tolerability in men with chemorefractory metastatic castration-resistant prostate cancer (CRPC).

SECONDARY OUTCOMES:
Evaluation of progression free survival | Every 9 weeks
  Preliminary evidence of durable efficacy will be based on a modified PCWG2-defined radiologic progression-free survival including RECIST 1.1 criteria (PFS).
Evaluation of overall response | Every 9 weeks
  Radiologic response criteria using RECIST 1.1 (overall response)
Preliminary evidence of response efficacy as measured by the rates of PSA decline (waterfall plot) and benchmarks of reaching a >30% decline within 3 months, a PSA decline >50% and >90%, and PSA normalization. Duration of PSA responses will be measured | Every 3 weeks
Favorable changes in circulating tumor cell number (5 or greater to less than 5) and proportion of men who achieve a reduction in CTC count | Every 3 weeks
Number and percent of participants that are alive | 2 years
  Overall survival
Detailed characterization of all NCI CTC v4.0 toxicities over time (per cycle) | Every 3 weeks
  Detailed characterization of all NCI CTC v4.0 toxicities over time (per cycle)
The concentration of tasquinimod and cabazitaxel in blood plasma | 12 weeks
  Pharmacokinetic analysis of tasquinimod and cabazitaxel (cycle 1-4 only)
Pain response, as measured by percentage of patients with a reduction of at least 2 points on the visual analog scale despite a stable pain regimen. Pain scores over time will be described in an exploratory fashion. | Every 3 weeks
Changes in bone alkaline phosphatase and LDH over time | Every 3 weeks
  Descriptive statistics will be used to summarize laboratory variables

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Armstrong, MD, Principal Investigator — Duke Cancer Institute
Locations (2):
- United States (2):
  - The University of Chicago, Chicago, Illinois
  - Duke Cancer Institute, Durham, North Carolina

REFERENCES:
- See also: Duke Cancer Institute — http://www.cancer.duke.edu